CLINICAL TRIAL: NCT04163549
Title: Evaluating the Effectiveness of the Safe at Home Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Rescue Committee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Safe at Home
Record Dates: First submitted 2019-11-12; First posted 2019-11-14 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2021-10

CONDITIONS: Family Functioning; Domestic Violence; Child Abuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Safe at Home Cycle 1 (Experimental): The experimental arm will receive the Safe at Home program which is a community-based discussion group series aiming to prevent and respond to intimate partner violence and child maltreatment in conflict-affected communities. It includes once weekly, single-sex discussion groups with coupled men and women and once monthly family discussion groups with couples and children. During the weekly sessions men and women reflect critically and engage in dialogue related to gender, power, and privilege, learn about the causes and consequence of violence against women and children and gain skills in stress management, psychosocial support and positive parenting strategies. Family sessions focus on improving relationship quality and shared decision-making among partners and participation of children in family decision-making.
  Interventions: Behavioral: Safe at Home
- Safe at Home Cycle 2 (No Intervention): During the period of the study, this group will not receive an intervention. Rather, this arm will receive the Safe at Home program after endline data collection is completed for a waitlisted group.

INTERVENTIONS:
Behavioral: Safe at Home — Discussion-based intervention
  Arms: Safe at Home Cycle 1

SUMMARY:
The goals of the pilot RCT examining the potential effectiveness of the Safe at Home program in DRC are to:

1. Determine the potential effectiveness of Safe at Home program on improvements of family functioning and secondary outcomes of reductions in intimate partner violence and child maltreatment
2. Determine the potential effectiveness of the Safe at Home program on changes in pathway outcomes such as attitudes towards harsh discipline, gender attitudes, power-sharing, positive parenting practices, etc.

DETAILED DESCRIPTION:
For the pilot RTC, quantitative data will be collected from up to 420 individuals participating in the Safe at Home program in the North Kivu, DRC. The 420 individuals comprising the study population will be 210 couples, of which both the male and female partners will be asked to participate in the study. After baseline data collection is completed, within each of the four sites where the program will occur in North Kivu, DRC, two groups of couples will be formed (n=8 groups total). Each group will be formed based on geographical proximity and will mirror real-life implementation of the program and ensure high fidelity to program design and limit contamination or spillover of Safe at Home to the control groups. Groups will then be randomized to receive Safe at Home in Cycle 1 or be waitlisted to receive Safe at Home in Cycle 2. After randomization is completed the Cycle 1 programming will commence. Following a waiting period of 3 months after the program ends, the endline survey will be administered. Subsequently Cycle 2 cohort will receive programming.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* registered for the Safe at Home program
* living with intimate partner who is also registered for the program and at least one child aged 6-12
* speaker of Swahili, Kinyarwanda, or French

Exclusion criteria includes:

* < 18 years of age
* being of a polygamous household
* not registered for program
* obvious mental, or cognitive, or communication difficulties.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 404 (Actual)
Dates: Start 2019-11-19 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2021-09-20 (Actual)

PRIMARY OUTCOMES:
Family functioning | Three months after intervention completion
  Mean change in women's reports (primary) and men's reports of family functioning

SECONDARY OUTCOMES:
Intimate partner violence | Three months after intervention completion
  Frequency change of past three month women's report of physical and/or sexual and/or emotional IPV (will also examine separately)
Harsh discipline | Three months after intervention completion
  Frequency change of past three month report of men's and women's physical or psychological harsh discipline practices against index child

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Falb, Principal Investigator — International Rescue Committee
Locations (1):
- International Rescue Committee, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Falb KL, Asghar K, Blackwell A, Baseme S, Nyanguba M, Roth D, Hategekimana JD. Improving family functioning and reducing violence in the home in North Kivu, Democratic Republic of Congo: a pilot cluster-randomised controlled trial of Safe at Home. BMJ Open. 2023 Mar 6;13(3):e065759. doi: 10.1136/bmjopen-2022-065759. PMID 36878658